CLINICAL TRIAL: NCT00714857
Title: Population Pharmacokinetics of Dexmedetomidine in ICU Patients
Acronym: Dex-Pop-PK
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Timo Iirola, MD, University of Turku
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: Dex-Pop-PK
Record Dates: First submitted 2008-07-07; First posted 2008-07-14 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Pharmacokinetics
Keywords: ICU patients; Dexmedetomidine; Sedation; Judged; Attending; Physician
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Patients receiving dexmedetomidine sedation
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — The patients are given a normal loading dose (10 min infusion at a rate of 3-6 μg/kg/h) of dexmedetomidine followed by continuous infusion of 0.1 - 2.5 μg/kg/h for the period of time the responsible physician finds reasonable.

SUMMARY:
Dexmedetomidine is a new, highly selective and potent alpha2-adrenoreceptor agonist registered for sedation of patients in intensive care units. Although the pharmacokinetics of dexmedetomidine have been studied previously also in an ICU setting, there is no information on the pharmacokinetics of long-lasting (>48 hours) dexmedetomidine infusions in humans.

The aim of this study is to study the pharmacokinetics of long-lasting dexmedetomidine infusions in ICU patients using the population pharmacokinetics approach.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Need for dexmedetomidine sedation (determined by the responsible physician).
* Predicted length of dexmedetomidine sedation ≥ 48 hours.
* Written informed consent from the patient or the relatives of the participating patient.

Exclusion Criteria:

* A previous history of intolerance to the study drug or related compounds and additives.
* Existing significant haematological, endocrine, metabolic or gastrointestinal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | Blood samples are taken three times daily for characterizing the pharmacokinetic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Timo T Iirola, M.D., Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland